CLINICAL TRIAL: NCT00483795
Title: Pilot Evaluation of Two Multipurpose Solutions in Regards to Corneal Staining
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 5308
Record Dates: First submitted 2007-06-01; First posted 2007-06-07 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Corneal Staining
MeSH Terms: interventions — Sodium Citrate; Sodium Chloride; sodium borate

INTERVENTIONS:
Drug: sodium citrate, sodium chloride, sodium borate, propylene glycol. citrate, tetronic 1304, AMP 95

SUMMARY:
To evaluate corneal staining after contact lens instillation with two different multi purpose solutions.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 yrs or older
* Males or females
* Any race or ethnic background
* CL patients using (multipurpose solutions) MPS
* Patients using Acuvue 2 lenses

Exclusion Criteria:

* Corneal refractive surgery within 6 months of this study.
* Contact lens use on day of examination.
* Corneal ectasia.
* Current use of Restasis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kislan, OD, Principal Investigator — Hazleton Eye Specialists
Locations (1):
- Hazleton Eye Specialists, Hazleton, Pennsylvania, United States